CLINICAL TRIAL: NCT05797662
Title: A Phase II Study of Propranolol for the Treatment of Kaposi Sarcoma in Children and Adults
Brief Title: A Study of Propranolol to Treat Kaposi Sarcoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-116; UM1CA121947 (NIH)
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Kaposi Sarcoma
Keywords: Kaposi Sarcoma; Propranolol
MeSH Terms: conditions — Sarcoma, Kaposi | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Propranolol (Experimental): Propranolol Twice Daily (BID) x 12 weeks Dosage: For ages ≤ 12 years: 3mg/kg/day divided BID; for ages > 12 years, 120 mg BID.
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — Adults: Propanolol 120 mg tablets by mouth twice daily for up to 24 weeks Children: Propanolol 3 mg/kg suspension, divided dose twice daily for up to 24 weeks

SUMMARY:
A clinical study of propranolol for the treatment of Kaposi Sarcoma in children and adults. This study will be an open-label single armed treatment trial that will test the effectiveness and the safety of treating Kaposi Sarcoma with propranolol.

DETAILED DESCRIPTION:
Eligible study participants will receive propanolol twice daily for an initial 12-week period. At the conclusion of 12-weeks, response will be assessed. Participants who achieve a complete or partial response will continue propanolol for an additional 6 weeks or 12 weeks, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric (< 18 years) and adult (≥ 18 years) participants with biopsy-proven and measurable Kaposi Sarcoma (KS) as defined in the KS Manual of Procedures (MOP).
* No urgent clinical indication for immediate cytotoxic chemotherapy. Participants who have received cytotoxic chemotherapy > 4 weeks prior to screening are eligible.
* KS stage:

  * < 18 years:

    * 1A (Mild): disease limited to skin, flat oral mucosal lesions, and/or flesh colored subcutaneous nodules, total <10 lesions.
    * 1B (Moderate): having any of the following features, alone or in combination: a total of 10-19 hyperpigmented skin/oral lesions, nodular oral involvement, conjunctival eye involvement, or exophytic mass.
  * ≥ 18 years:

    * T0: confined to skin and/or lymph nodes and/or minimal oral lesions.
    * T1: limited to tumor-associated edema of cutaneous lesions without functional impairment or flat oral lesions.
* Performance Status:

  * < 18 years:

    * Lansky performance status > 70%
  * ≥ 18 years:

    * Easter Cooperative Oncology Group (ECOG) performance status ≤ 2
* Participants must have adequate organ function, as defined by the following:

  * Bilirubin (direct or total) within normal range, or total bilirubin <3.0 mg/dl for participants with Gilbert syndrome.
  * Calculated creatinine clearance ≥ 30 mL/min for participants ≥ 12 years (see Appendix III); creatinine <1.5 Upper Limit Normal (ULN) for participants < 12 years.
  * Hemoglobin > 9 g/dL;
  * Platelets > 100 × 109/L;
  * ANC > 1000 cells/mm3
* Human Immunodeficiency Virus (HIV) positive participants must be on antiretroviral therapy (ART) that conforms to local standards of care. Participants will have been on ART for at least 12 weeks. Participants will not be excluded based on CD4 count or HIV viral load.
* HIV positive participants must not show recent improvement on ART that may confound response evaluation:

  * If on ART 12 to 24 weeks, participants must show evidence of KS progression requiring further systemic treatment.
  * If on ART for >24 weeks, must show no evidence of regression in the last eight weeks.
* HIV-negative participants must not show evidence of improvement in the three months prior to enrollment.
* No history of asthma or diabetes mellitus (as it is a risk factor for hypoglycemia).
* No clinically significant cardiovascular disease other than hypertension, which is permitted.
* No use of beta-adrenergic antagonists for other indications.
* Not pregnant or planning to become pregnant. Propranolol is United Stats Food and Drug Administration (US FDA) pregnancy category C. At this time, the study team has determined that the unknown risk to a developing fetus is greater than the potential benefit of treatment.
* Use of effective contraception for women of childbearing potential, defined as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months.
* Women of child bearing potential (WOCBP) must agree to use adequate contraception (oral contraceptive pills, intrauterine device, Nexplanon, Depo-Provera, or permanent sterilization, etc., or another acceptable method as determined by the investigator) prior to study entry, for the duration of study participation.
* Not breast feeding.

Exclusion Criteria:

• Participants who do not fulfill the criteria as listed in Section 3.1 above, are ineligible. Additionally, the presence of any of the following conditions will exclude a participant from study enrollment:

* Children and adolescents with lymph node or visceral disease, woody edema, or ≥ 20 cutaneous lesions.
* Children and adolescents with heart rate or systolic blood pressure <10th percentile for age.
* Adults with visceral disease or tumor-associated edema causing functional impairment.
* Shortness of breath, hemoptysis, or moderate/severe cough not attributable to causes other than KS.
* Bleeding from the mouth or rectum not attributable to causes other than KS.
* Treatment for active and serious infection.
* Children with severe acute malnutrition based on World Health Organization (WHO) criteria (Mid-upper arm circumference <11.5 cm, weight-for height Z-score <-3 or presence of symmetrical pitting edema).
* Given the risk of hypotension and hypoglycemia, participants must take the study drug with food. If needed, the study team will pursue additional funding to support providing supplemental food for participants who experience food insecurity.
* Patients who experienced hypersensitivity to propranolol during initiation phase of treatment or had previous known allergy to propranolol or allergy to other β-blockers.
* Patients with a history of uncompensated heart failure; severe sinus bradycardia; sick sinus syndrome; or heart block greater than first-degree.
* Patients with diagnosed obstructive airway disease such as asthma, chronic obstructive pulmonary disease (COPD), or bronchiolitis.
* History of diabetes mellitus (as it is a risk factor for hypoglycemia)
* Patients receiving concurrent treatment with an anticancer therapy. Patients must not have received any anticancer therapies within 30 days prior to receiving the first dose of investigational treatment.
* Patients with concern for Kaposi Sarcoma herpesvirus (KSHV) inflammatory cytokine syndrome.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | At one year
  ORR is defined as the proportion of participants with complete response (CR), or partial response (PR) based on AIDS Malignancy Consortium Kaposi Sarcoma (AMC KS) Response Criteria.

SECONDARY OUTCOMES:
Number of dose-limiting toxicities | At one year
  To evaluate the number of dose-limiting toxicities. The dose-limiting toxicities will be based on the National Cancer Institute's Common Terminology Criteria for Adverse Events
Number of treatment-emergent adverse events | At one year
  To evaluate the number of treatment-emergent adverse events. The treatment-emergent adverse events will be based on the National Cancer Institute's Common Terminology Criteria for Adverse Events
Complete and Partial Response rates in children and adults | At one year
  Proportion of children and adults with a Complete Response or Partial Response.
Time to recurrence among children | At one year
  Time to recurrence among responders overall in children. Recurrent disease is defined as the appearance of tumor following documentation of a complete remission.
Time to recurrence among adults | At one year
  Time to recurrence among responders overall in adults. Recurrent disease is defined as the appearance of tumor following documentation of a complete remission.
Time to progression among children | At one year
  Time to progression among responders overall in children. Time to progression is defined as time from initiation of propranolol to documentation of first progression.
Time to progression among adults | At one year
  Time to progression among responders overall in adults. Time to progression is defined as time from initiation of propranolol to documentation of first progression.

CONTACTS AND LOCATIONS:
Overall Officials: Shane McAllister, Md, PhD, Study Chair — University of Minnesota Medical School Department of Pediatrics
Locations (9):
- Fundación Huésped, Buenos Aires, Argentina
- Brazil (2):
  - Instituto Nacional de Câncer José de Alencar, Rio de Janeiro
  - Complexo Hospitalar Universitário Professor Edgard Santos, Salvador
- Moi University School of Medicine, Eldoret, Kenya
- UNC Project Malawi, Lilongwe, Malawi
- Instituto Nacional de Cancerologia, Mexico City, Mexico
- African Cancer Institute at Stellenbosch, Cape Town, South Africa
- Uganda Cancer Institute, Kampala, Uganda
- University of Zimbabwe College of Health Sciences, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Undecided